CLINICAL TRIAL: NCT05881265
Title: Multi-center Phase II Prospective Study for the Treatment of Chidamide and Venetoclax in Patients With All-trans Retinoic Acid (ATRA) and Arsenic (As) Resistant Acute Promyelocytic Leukemia (APL)
Brief Title: Treatment of Chidamide and Venetoclax for Retinoic Acid and Arsenic Resistant Acute Promyelocytic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Clinical Research Center (Unknown)
Responsible Party: Principal Investigator, Jiong HU, Head, Blood & Marrow Transplantation Center, Rui Jin Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R/R-APL-2023
Record Dates: First submitted 2023-05-16; First posted 2023-05-31 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: APL
Keywords: refractory，APL

STUDY DESIGN:
Intervention Model Description: Chi-Ven treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chi-Ven treatment (Experimental): Patients receive chidamide and venetoclax treatment
  Interventions: Drug: Chidamide+venetoclax

INTERVENTIONS:
Drug: Chidamide+venetoclax — Chidamide 30mg BIW x 4 weeks; Venetoclax 100mg D1, 200mg D2 and 400mg D3-28
  Other Names: Chi-VEN

SUMMARY:
Based on the current treatment with retinoic acid (ATRA) and arsenic (As), most patients with APL achieved long-term survival. There are few patients relapsed and became refractory to the RA and As treatment. In our pre-clinical study, we found that targeting histone deacetylase inhibitor 3 (HDAC3)degraded PML-RARa oncoprotein and induced differentiation and apoptosis of RA and As resistant APL in vitro and in vivo. In this study, we evaluate the efficacy and feasibility of combination therapy for HDAC3 inhibitor and venetoclax in patients with refractory APL.

DETAILED DESCRIPTION:
For patients with newly-diagnosed acute promyelocytic leukemia (APL), the combination therapy retinoic acid (ATRA) combined with arsenic (As) is the mainstay upfront treatment. Most patients enjoy long-term survival with or without chemotherapy. Even though with such good prognosis, there are still some patients relapsed and eventually became refractory to RA and As treatment. In our pre-clinical study, we demonstrate that targeting histone deacetylase inhibitor 3 (HDAC3) could degrade PML-RARa oncoprotein and induce differentiation and apoptosis of RA and As resistant APL in vitro and in vivo. In this multi-center prospective study, we evaluate the efficacy and feasibility of combination therapy for HDAC3 inhibitor (chidamide) and venetoclax in patients with refractory APL.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PML-RARα+ APL
* Patients in non-remission status after treatment of RA combined with As
* Patients with life expectance >=3 months
* Inform consent provided

Exclusion Criteria:

* Patients with incontrollable infection
* Patients with life-expectancy less than 2 months
* Patients with abnormal liver (>3XN) and renal function (>3XN）

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
complete remission and complete remission with incomplete recovery of peripheral blood count | Day 42
  patients with <5% promyelocytes in bone marrow with or without full recovery of peripheral cell count

SECONDARY OUTCOMES:
Overall survival | 1 year
  Patients alive
Leukemia-free survival | 1 year
  Patients alive without leukemia relapse
Non-relapse mortality | 1 year
  Patients died without documentation of leukemia relapse
relapse | 1 year
  Patients with documentation of leukemia relapse
Early death | 42 days
  Patients died of any causes

CONTACTS AND LOCATIONS:
Overall Officials: Chun Wang, Study Director — Zhaxin Hospital, Go Broad Health Care
Locations (5):
- China (5):
  - The Affiliated Huai An No 1 Perople's Hospital of NanJing University, Huai'an, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jiong HU, Shanghai, Shanghai Municipality
  - Zhaxin Hospital, Go Broad Health Care, Shanghai, Shanghai Municipality
  - NanFang Hospital, Guangzhou

IPD SHARING:
Plan to Share IPD: No
Individual participant data is available only based on request to study director or principle investigator